CLINICAL TRIAL: NCT03157869
Title: Influence of Transcranial Direct Stimulation Current on Motor Learning of Young Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Maria Elisa Pimentel Piemonte, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: tDCS1
Record Dates: First submitted 2017-05-01; First posted 2017-05-17 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Learning, Automatism, Motor Activity, Electric Stimulation
MeSH Terms: conditions — Motor Activity | interventions — Transcranial Direct Current Stimulation; Simulate composite resin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Direct Current Stimulation (Experimental): * Intervention: anodic tDCS (20 minutes ON, intensity 2milliamps) on the primary motor cortex contralateral of the trained hand (right) simultaneously to the motor training and supraorbital cathode ipsilateral
  * Motor training will consist of 8 blocks with 300 repetitions of sequential finger movements performed with the right hand.
  Interventions: Device: Transcranial Direct Current Stimulation
- Control (Sham Comparator): * Intervention: simulated anodic tDCS (30 seconds ON, intensity 2milliamps) on the primary motor cortex contralateral of the trained hand (right) simultaneously to the motor training and supraorbital cathode ipsilateral
  * Motor training will consist of 8 blocks with 300 repetitions of sequential finger movements performed with the right hand.
  Interventions: Other: Simulated

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Anodic tDCS during 20 minutes ON, intensity 2milliamps, on the contralateral motor cortex of the trained hand simultaneously with the motor training. The cathode (negative electrode) will be positioned over the contralateral supraorbital region. It wil be used rubber electrodes covered by a vegetal electrode embedded in saline solution, physiological saline, measuring 5 x 5 cm (25 cm2).
  Arms: Transcranial Direct Current Stimulation
Other: Simulated — Simulated anodic tDCS (only 30 seconds ON), intensity 2milliamps, on the contralateral motor cortex of the trained hand simultaneously with the motor training. The cathode (negative electrode) will be positioned over the contralateral supraorbital region. It wil be used rubber electrodes covered by a vegetal electrode embedded in saline solution, physiological saline, measuring 5 x 5 cm (25 cm2).
  Arms: Control

SUMMARY:
Motor learning occurs with structural and functional modifications in neural networks that meet a certain demand. The improvement of performance in diverse activities is a measure of learning, as well as the generalization and transference of this capacity. Transcranial direct current stimulation (tDCS) is a modulation technique of brain activity that modifies cortical excitability, causing changes in motor evoked potentials that influence motor learning. Modifications similar to the long-term potentiation, essential for learning processes, have also been described after applying tDCS. The primary motor cortex is the area of stimulation where there is more robust evidence in favor of increased motor learning. PURPOSE: to investigate the effects of anodic tDCS on the learning of sequential finger movements in young and healthy individuals.

DETAILED DESCRIPTION:
Thirty-six young healthy individuals, right-handed, with no deficits that difficult the performance of the procedures will participate in the study. These individuals will be randomly divided into an experimental group that will perform the motor training of a sequential task of fingers simultaneously to the anodic tDCS on the contralateral motor cortex the trained hand and a control group that will perform the same training simultaneously the stimulation placebo (simulated in the same region of the experimental group). The training will consist of 8 blocks with 300 repetitions of sequential finger movements performed with only the right upper limb. The speed and accuracy of sequential movements will be used as a measure of performance. These measures will be performed prior to training, immediately after, 48 hours, 7 days, and 28 days after trained hand training (TH) for assessment of short and long term learning. In addition, performance evaluations (1) of the reverse-trained sequence in TH will be performed to evaluate the generalization; (2) of the trained sequence in left hand (non-trained) to evaluate the intermanual transfer; and (3) trained sequence in TH in double-task condition to evaluate automaticity. Appropriate statistical methods will be used to identify inter- and intra-group differences.

ELIGIBILITY:
Inclusion Criteria:

* Young subjects aged between 18 and 35 years, right-hand (evaluated by the Edinburgh Inventory), of both genders, attending the third grade in a private university.

Exclusion Criteria:

* Individuals using central nervous system drugs with uncorrected visual and / or auditory disorders who have any neurological, psychiatric, or orthopedic diseases and who have differentiated finger, musician or typist skills will be excluded.

Due to the electrostimulation procedure, individuals who use hair chemistry, individuals who have a metallic implant on the head or a pacemaker, and who have scars in the region to be stimulated will also be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-11-05 (Estimated)

PRIMARY OUTCOMES:
Speed | Up to 28 days
  The speed (number of repetitions in a minute) of sequential movements will be used as a measure of performance. These measures will be performed prior to training, immediately after, 48 hours, 7 days, and 28 days after trained hand training (TH) for assessment of short and long term learning. In addition, performance evaluations (1) of the reverse-trained sequence in TH will be performed to evaluate the generalization; (2) of the trained sequence in left hand (non-trained) to evaluate the intermanual transfer; and (3) trained sequence in TH in double-task condition to evaluate automaticity.
Accuracy | Up to 28 days
  The accuracy (number of errors in a minute) in the same way as described to Outcome 1

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PhD, Study Director — University of Sao Paulo
Locations (1):
- Center of Research of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No